CLINICAL TRIAL: NCT01930734
Title: Randomized-Controlled-Double Blind Trial of Low Dose Dobutamine in Advanced Heart Failure Patients in a Day-Care Clinic
Brief Title: Outcome and Safety of Intermittent Dobutamine Infusion at a Day-Care Center in Advanced Heart Failure Patients
Acronym: DoBHF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-13-0341-DF-CTIL
Record Dates: First submitted 2013-08-25; First posted 2013-08-29 (Estimated); Last update posted 2013-08-30 (Estimated); Status verified 2013-08

CONDITIONS: Heart Failure
Keywords: Heart Failure; Dobutamine
MeSH Terms: conditions — Heart Failure | interventions — Dobutamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal Saline (Placebo Comparator): Normal Saline Placebo infusion containing Normal Saline NaCl 0.9% twice a week for a total duration of 6 months.
  Placebo will be given at the same rate as the Dobutamine infusion, under the same measures.
  Interventions: Drug: Normal Saline
- Dobutamine (Experimental): Twice weekly, IV Dobutamine infusion up to 5mcg/Kg/min infusion, for the duration of 6 months. Medication will be administered under medical supervision and continues ECG and vital sign monitoring. Routine electrolyte and renal function testing will be performed and electrolytes corrected as indicated.
  Interventions: Drug: Dobutamine

INTERVENTIONS:
Drug: Dobutamine — Dobutamine infusion up to 5mcg/Kg/min
  Other Names: Dobutrex
  Arms: Dobutamine
Drug: Normal Saline — Normal Saline solution 0.9% Placebo Arm
  Arms: Normal Saline

SUMMARY:
Heart failure (HF) is a prevalent disease reaching 1-2% of adult population in developed countries, and 10% in patients over 70 years. In the past HF patients had a 5-year mortality rate of 60-70% of HF with high rate of hospitalization and disability leading to a HF epidemic. Treatment improvements in the past decades have significantly reduced hospitalization and mortality. However, there is an increasing subset of patients (>10%) with advanced HF symptoms (functional class III/IV) for whom current management strategies are limited and do not provide a significant improvement in morbidity, mortality and quality of life.

Specialized HF clinics, implementing a comprehensive therapeutic approach, were suggested to be beneficial in this population. However, the design of these clinics is variable with different methods of follow-up, therapy and supervision. Intermittent infusions of dobutamine were previously inconclusive regarding symptom alleviation and hemodynamic improvement and raised a concern of increased mortality in HF patients. Furthermore, the evidence scope is narrow since most trials including inconsistent and relatively high dobutamine dosages. Accordingly, current guidelines do not provide specific recommendations for dobutamine therapy in stable HF patients, and indication for treatment are limited for acute HF with hypotension and signs of hypoperfusion, or alleviation of symptoms in severely symptomatic patients in stage D HF.

The primary aim of the proposed study is to evaluate the impact of intermittent low-dose dobutamine infusion on clinical and hemodynamic parameters in advanced HF patients treated in a tertiary heart failure clinic in the setting of a randomized clinical trial. We hypothesize that intermittent therapy with low-dose dobutamine will be associated with improved functional capacity and quality of life among patients with advanced heart failure, thereby providing evidence for beneficial effects of a potentially important therapeutic regimen in this high risk population.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Symptomatic HF with NYHA III-IV
* Left ventricular ejection fraction < 30%
* Maximal tolerated dosage of Angiotensin receptor blocker (ARB) or Angiotensin converting enzyme inhibitor (ACEI), aldosterone antagonists and β-Blockers according to blood pressure, heart rate, renal function and potassium levels
* Prior implementation of resynchronization therapy and implantable defibrillator as indicated??
* Prior HF hospitalization in the past 12 months
* Unsatisfactory response to intravenous diuretics during hospitalization or ambulatory care.

Exclusion Criteria:

* Active ischemia
* Acute coronary syndrome or cardiac surgery within 3 months
* Hemodynamic and respiratory instability, with systolic blood pressure below 85mmHg, and oxygen saturation below 90% at rest
* Uncontrolled hypertension >180/110 mmHg
* Contra-indication to dobutamine therapy
* Hemodialysis therapy
* Malignant ventricular arrythmias
* Drug or alcohol abuse
* Sepsis or ongoing systemic infection
* Active myocarditis
* Severe valvular stenosis
* Non-compliance
* Life-threatening extra-cardiac disease or malignancy with a life expectancy below 1 year
* Inability to sign an informed consent
* Participation in another trial during the previous 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
• Improvement in maximal oxygen consumption (VO2 max) | 6 months and 12 months

SECONDARY OUTCOMES:
• Combined endpoint of heart failure or all-cause mortality at 6 and 12 months of follow-up | 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Dov Freimark, Prof. MD., Principal Investigator — Leviev Heart Center
Locations (1):
- Leviev Heart Center, Chaim Sheba Medical Center, Ramat Gan, Israel